CLINICAL TRIAL: NCT01602614
Title: Evaluation of the Pharmacokinetics and Pharmacodynamics of Ganciclovir in Premature Infants Receiving Treatment for Cytomegalovirus Infection
Brief Title: Evaluation of the Pharmacokinetics (PK) and Pharmacodymamics (PD) of Ganciclovir (GCV) in Premature Infants Receiving Treatment for Cytomegalorivus (CMV) Infection
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Kimberlin, MD, Protocol Principal and Lead Investigator, University of Alabama at Birmingham
Other Study IDs: F21116007
Record Dates: First submitted 2012-05-17; First posted 2012-05-21 (Estimated); Results first posted 2020-05-19 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Remnant blood will be retained for future cytomegalovirus (CMV) studies if subjects/subject families consent to future use. Institutional Review Board (IRB) approval for any future studies of remnant specimens will be required.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group 1: ≤ 27 weeks 6 days gestational age at birth and ≤ 30 days chronologic age at study enrollment. Dose and duration of intravenous ganciclovir therapy is at the discretion of the treating physician and will not be dictated by the research protocol.
- Group 2: ≤ 27 weeks 6 days gestational age at birth and > 30 days chronologic age at study enrollment. Dose and duration of intravenous ganciclovir therapy is at the discretion of the treating physician and will not be dictated by the research protocol.
- Group 3: ≥ 28 weeks 0 days gestational age at birth and ≤ 30 days chronologic age at study enrollment. Dose and duration of intravenous ganciclovir therapy is at the discretion of the treating physician and will not be dictated by the research protocol.
- Group 4: ≥ 28 weeks 0 days gestational age at birth and > 30 days chronologic age at study enrollment. Dose and duration of intravenous ganciclovir therapy is at the discretion of the treating physician and will not be dictated by the research protocol.

SUMMARY:
This is a clinical sampling study, and no study drugs will be administered under this protocol. Premature infants who receive intravenous ganciclovir as part of clinical care will be eligible for participation in this study. Intravenous ganciclovir will not be provided under this protocol.

DETAILED DESCRIPTION:
This is an open-label, multi-center, clinical sampling study to assess ganciclovir pharmacokinetics and pharmacodynamics in premature infants. Only those subjects who receive ganciclovir for clinical reasons will be enrolled. The decision to initiate ganciclovir therapy will be made by the attending physician based upon his/her clinical decision to treat virologically-confirmed CMV infection; infants receiving such therapy and meeting entry criteria will then be eligible for this study. Therefore, ganciclovir will not provided under this protocol.

Subjects meeting enrollment criteria will be entered into this clinical trial. Subjects will be stratified by gestational age and by chronologic age as follows: 1) ≤ 27 weeks 6 days gestational age at birth and ≤ 30 days chronologic age at study enrollment; 2) ≤ 27 weeks 6 days gestational age at birth and > 30 days chronologic age at study enrollment; 3) ≥ 28 weeks 0 days gestational age at birth and ≤ 30 days chronologic age at study enrollment; 4) ≥ 28 weeks 0 days gestational age at birth and > 30 days chronologic age at study enrollment. Eight subjects will enroll in each of the four groups, for a total sample size of 32 subjects. Subjects in each cohort with inadequate pharmacokinetic data for analysis (e.g., due to dropping out of the study before PK assessments are performed, or blood sampling obtained but is inadequate for analysis) will be replaced and will not count toward the total of eight subjects in each of the four groups. Additionally, enrollment of an additional 2-3 subjects may be allowed for operational reasons.

A full pharmacokinetic profile will be obtained with one of the ganciclovir doses received after enrollment. PK assessments will be obtained after the subject has received study assessment dose 3, 4, 5, 6, 7, or 8 of intravenous ganciclovir. Specimens will be shipped for processing at that time. The pharmacokinetic data will then be provided to the study site, including the area under curve (AUC) and clearance (CL) values for information purposes.

Duration of intravenous ganciclovir therapy is at the discretion of the treating physician and will not be dictated by the research protocol. Both whole blood for CMV polymerase chain reaction (PCR) and urine for CMV detection will be obtained once in each study period as long as the subject is receiving intravenous ganciclovir therapy. These specimens will be used to determine blood viral load and ganciclovir resistance. Since ganciclovir is a renally excreted drug, serum creatinine will be drawn for the research protocol on the day that the ganciclovir pharmacokinetic specimens are obtained in order to calculate creatinine clearance using a method such as the modified Schwartz formula, and thus correlate ganciclovir clearance with renal function. Otherwise, data from hematology assessments (WBC count and differential, hemoglobin, platelet count) and from chemistry labs (serum creatinine, aspartate aminotransferase (AST) , and alanine aminotransferase (ALT) will be recorded on the study case report forms during each study period if they are being obtained for clinical reasons, but will not be drawn only for the purposes of the study. Ganciclovir dosing information (mg/dose, dosing interval, and patient weight) will be recorded on the day of the pharmacokinetic blood draws, and weekly from Period 1 through Period 7 as long as the subject is receiving intravenous ganciclovir therapy.

If the patient continues to receive intravenous ganciclovir from Study Assessment Day 18 through Study Assessment Day 24 (Period 4), a second PK assessment may be performed at the request of the treating physician if the subject weighs 575 grams or more at the time of specimen collection.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent from parent(s) or legal guardian(s)
2. Confirmation of CMV infection from urine, blood, or saliva by culture, shell vial, or PCR tests (local lab)
3. Receiving intravenous ganciclovir, prescribed by the patient's physician
4. < 32 weeks gestational age at birth
5. ≥ 500 grams at study enrollment

Exclusion Criteria:

1. Imminent demise
2. Current receipt of valganciclovir or foscarnet
3. Receiving breast milk from a mother who is being treated with ganciclovir or valganciclovir
4. Current receipt of other investigational drugs
5. Major congenital anomaly that in the site investigator's opinion may impact drug metabolism or the patient's volume of distribution

Ages: 1 Day to 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants who receive intravenous ganciclovir as part of clinical care
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-04; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Kimberlin, MD, Principal Investigator — University of Birmingham at Alabama; Richard Whitley, MD, Principal Investigator — University of Alabama at Birmingham
Locations (15):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of South Florida School of Medicine, St. Petersburg, Florida
  - Louisiana State University Health Science Center - Shreveport, Shreveport, Louisiana
  - Johns Hopkins Medical Institutions, Baltimore, Maryland
  - Washington University in St Louis School of Medicine, St Louis, Missouri
  - Steven & Alexandra Cohen Children's Medical Center of New York (CCMC), Manhasset, New York
  - University of Rochester, Rochester, New York
  - Carolinas Medical Center - Charlotte, Charlotte, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Nationwide Childrens Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 0 | 10 | 8 | 0
Completed | 0 | 10 | 8 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Group 1 and Group 4 did not enroll subjects.
Groups:
- Group 1: ≤ 27 weeks 6 days gestational age at birth and ≤ 30 days chronologic age at study enrollment
- Group 2: ≤ 27 weeks 6 days gestational age at birth and > 30 days chronologic age at study enrollment
- Group 3: ≥ 28 weeks 0 days gestational age at birth and ≤ 30 days chronologic age at study enrollment
- Group 4: ≥ 28 weeks 0 days gestational age at birth and > 30 days chronologic age at study enrollment
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 0 | 10 | 8 | 0 | 18
Age, Customized [Mean (Standard Deviation); unit: days]
  Age (days) |  | 63.2 (18.0) | 16.5 (7.4) |  | 42.4 (27.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 2 | 1 |  | 3
  Male |  | 8 | 7 |  | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian |  | 1 | 0 |  | 1
  Race: Black or African American |  | 3 | 0 |  | 3
  Race: White |  | 5 | 7 |  | 12
  Race: More than one race |  | 1 | 1 |  | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  | 10 | 8 |  | 18

OUTCOME MEASURES:

1. Primary Outcome: Plasma Pharmacokinetics Parameters for Ganciclovir Area Under the Curve at 12 Hours (AUC12mgxh/L)
Description: A series of blood samples will be collected to assess the ganciclovir levels in the blood at the following time points: 0 hour (immediately prior to intravenous (IV) ganciclovir dose; within 15 min prior to dose), 1 hour (immediately after the end of the IV ganciclovir dose; within 15 min after dose), 2-3 hour, 5-7 hour, and 10-12 hour; required amount of whole blood for plasma ganciclovir determination at each time point is at least 0.2 mL
Time Frame: within 12 hours after dose administration
Population: No subjects were enrolled in Group 1 and Group 4. One subject in Group 3 did not collect full panel therefore no pk analyzed.
Measure: Mean (Standard Error); unit: mgxh/L
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 0 | 10 | 7 | 0
mgxh/L |  | 47.2 (21.5) | 76.8 (39.6) |

2. Secondary Outcome: Plasma Pharmacokinetics Parameters for Ganciclovir, Including Maximum Serum Concentration (Cmax mg/L).
Description: Looking at the Pharmacokinetics (PK) parameters for Ganciclovir (GCV). A series of blood samples was collected to assess the ganciclovir levels in the blood at the following time points: 0 hour (immediately prior to intravenous (IV) ganciclovir dose; within 15 min prior to dose), 1 hour (immediately after the end of the IV ganciclovir dose; within 15 min after dose), 2-3 hour, 5-7 hour, and 10-12 hour.
Time Frame: within 12 hours after dose administration
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 0 | 10 | 7 | 0
mg/L |  | 7.9 (2.2) | 10.0 (5.4) |

3. Secondary Outcome: Plasma Pharmacokinetics Parameters for Ganciclovir for Half-life (T1/2 hr).
Description: as for outcome 2
Time Frame: within 12 hours after dose administration
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Hr
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 0 | 10 | 7 | 0
Hr |  | 5.0 (3.5) | 7.2 (2.2) |

4. Secondary Outcome: Plasma Pharmacokinetics Parameters for Ganciclovir for Clearance (Cl L/hr/kg).
Description: as for outcome 2
Time Frame: within 12 hours after dose administration
Population: as for outcome 1
Measure: Mean (Standard Error); unit: L/hr/kg
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 0 | 10 | 7 | 0
L/hr/kg |  | 0.1 (0.1) | 0.1 (0.0) |

5. Secondary Outcome: Plasma Pharmacokinetics Parameters for Ganciclovir for Volume of Distribution (Vd L).
Description: as for outcome 2
Time Frame: within 12 hours after dose administration
Population: as for outcome 1
Measure: Mean (Standard Error); unit: L
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 0 | 10 | 7 | 0
L |  | 1.4 (0.6) | 1.1 (0.3) |

6. Secondary Outcome: Correlation of Ganciclovir Plasma Pharmacokinetics (Clearance (CL) With Whole Blood Cytomegalovirus (CMV) Viral Load.
Description: Comparing the GCV PK clearance (CL L/hr/kg) results to the whole blood CMV viral load data.
Time Frame: 6 weeks
Population: No subjects were enrolled in Group 1 and Group 4. Four (4) Group 2 subjects and two (2) Group 3 subjects did not have viral loads for at least two (2) time points, therefore correlation could not be performed.
Measure: Mean (Standard Deviation); unit: L/hr/kg
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 0 | 6 | 6 | 0
L/hr/kg |  | 0.13667 (0.08311) | 0.08000 (0.02530) |
Statistical Analysis 1: Comparison: Group 2 vs Group 3; No subjects were enrolled in Group 1 and Group 4. One subject in Group 3 did not collect full PK panel therefore no pk was analyzed for this subject; Test type: Other — Spearman Rank Correlation; p = 0.3117, Spearman Rank Correlation

7. Secondary Outcome: Correlation of Ganciclovir Plasma Pharmacokinetics Maximum Serum Concentration (Cmax) With Whole Blood Cytomegalovirus (CMV) Viral Load.
Description: Comparing the GCV PK results maximum serum concentration (Cmax) to the CMV viral load data.
Time Frame: 6 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 0 | 6 | 6 | 0
mg/L |  | 7.99833 (2.78494) | 10.22500 (5.82284) |
Statistical Analysis 1: Comparison: Group 2 vs Group 3; [analysis description as in outcome 6, analysis 1]; Test type: Other — Spearman Rank Correlation; p = 0.6175, Spearman Rank Correlation — Spearman Rank Correlation

8. Secondary Outcome: Correlation of Ganciclovir Plasma Pharmacokinetics Area Under the Curve (AUC12) With Whole Blood Cytomegalovirus (CMV) Viral Load.
Description: Comparing the GCV PK results area under the curve (AUC12-mgxh/L) to the whole blood CMV viral load data.
Time Frame: 6 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mgxh/L
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 0 | 6 | 6 | 0
mgxh/L |  | 50.77167 (26.46657) | 79.58833 (42.67824) |
Statistical Analysis 1: Comparison: Group 2 vs Group 3; [analysis description as in outcome 6, analysis 1]; Test type: Other — Spearman Rank Correlation; p = 0.7129, Spearman Rank Correlation — Spearman Rank Correlation

9. Secondary Outcome: Correlation of Ganciclovir Plasma Pharmacokinetics Half-life (T1/2) With Whole Blood Cytomegalovirus (CMV) Viral Load.
Description: Comparing the GCV PK results half-life (T1/2 hr) to the whole blood CMV viral load data.
Time Frame: 6 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 0 | 6 | 6 | 0
hr |  | 5.37333 (4.34650) | 7.36167 (2.39133) |
Statistical Analysis 1: Comparison: Group 2 vs Group 3; [analysis description as in outcome 6, analysis 1]; Test type: Other — Spearman Rank Correlation; p = 0.9828, Spearman Rank Correlation

10. Secondary Outcome: Correlation of Ganciclovir Plasma Pharmacokinetics Volume of Distribution (Vd) With Whole Blood Cytomegalovirus (CMV) Viral Load.
Description: Comparing the GCV PK results volume of distribution (Vd L) to the whole blood CMV viral load data.
Time Frame: 6 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 0 | 6 | 6 | 0
L |  | 1.36333 (0.74457) | 1.06000 (0.35491) |
Statistical Analysis 1: Comparison: Group 2 vs Group 3; [analysis description as in outcome 6, analysis 1]; Test type: Other — Spearman Rank Correlation; p = 0.9656, Spearman Rank Correlation

11. Secondary Outcome: Correlation of Ganciclovir Plasma Pharmacokinetics Clearance (Cl) With Clearance of CMV in Urine
Description: Comparing the GCV PK results clearance (Cl L/hr/kg) to the clearance of CMV in the urine samples
Time Frame: 6 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L/hr/kg
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 0 | 6 | 6 | 0
L/hr/kg |  | 0.12000 (0.08025) | 0.07667 (0.02160) |
Statistical Analysis 1: Comparison: Group 2 vs Group 3; [analysis description as in outcome 6, analysis 1]; Test type: Other — Spearman Rank Correlation; p = 0.5113, Spearman Rank Correlation

12. Secondary Outcome: Correlation of Ganciclovir Plasma Pharmacokinetics Maximum Serum Concentration (Cmax) With Clearance of CMV in Urine.
Description: Comparing the GCV PK results to the Cmax with clearance of CMV in the urine samples
Time Frame: 6 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 0 | 6 | 6 | 0
mg/L |  | 8.93000 (1.91465) | 10.58667 (5.58772) |
Statistical Analysis 1: Comparison: Group 2 vs Group 3; [analysis description as in outcome 6, analysis 1]; Test type: Other — Spearman Rank Correlation; p = 0.2170, Spearman Rank Correlation — Spearman Rank Correlation

13. Secondary Outcome: Correlation of Ganciclovir Plasma Pharmacokinetics Area Under the Curve (AUC) With Clearance of CMV in Urine.
Description: Comparing the GCV PK AUC results to the clearance of CMV in the urine samples.
Time Frame: 6 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mgxhr/L
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 0 | 6 | 6 | 0
mgxhr/L |  | 55.23667 (23.90314) | 81.46333 (41.29835) |
Statistical Analysis 1: Comparison: Group 2 vs Group 3; [analysis description as in outcome 6, analysis 1]; Test type: Other — Spearman Rank Correlation; p = 0.4299, Spearman Rank Correlation — Spearman Rank Correlation

14. Secondary Outcome: Correlation of Ganciclovir Plasma Pharmacokinetics Maximum Serum Half Life (T1/2) With Clearance of CMV in Urine.
Description: Comparing the GCV PK half-life results to the clearance of CMV in the urine samples.
Time Frame: 6 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 0 | 6 | 6 | 0
hr |  | 6.25000 (4.04001) | 7.39667 (2.36849) |
Statistical Analysis 1: Comparison: Group 2 vs Group 3; [analysis description as in outcome 6, analysis 1]; Test type: Other — Spearman Rank Correlation; p = 0.8629, Spearman Rank Correlation — Spearman Rank Correlation

15. Secondary Outcome: Correlation of Ganciclovir Plasma Pharmacokinetics Volume of Distribution (Vd) With Clearance of CMV in Urine.
Description: Comparing the GCV PK Vd results to the clearance of CMV in the urine samples
Time Frame: 6 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 0 | 6 | 6 | 0
L |  | 1.35000 (0.74814) | 0.97333 (0.25073) |
Statistical Analysis 1: Comparison: Group 2 vs Group 3; [analysis description as in outcome 6, analysis 1]; Test type: Other — Spearman Rank Correlation; p = 0.5717, Spearman Rank Correlation — Spearman Rank Correlation

ADVERSE EVENTS:
Time Frame: Adverse events were observed during the 42 day study period.
Description: * Adverse Events (AEs) associated with blood draws
  * All adverse events that meet the reporting requirements of the Institutional Review Board (which will also be reported to Protocol Chair, Division of Microbiology and Infectious Diseases (DMID) Medical Officer, Medical Monitor and the Clinical Project Manager).
  All Adverse Events (AEs) as described above will be followed until resolved or considered stable.
  No adverse events were reported.
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/10 | 0/8 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/10 | 0/8 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/10 | 0/8 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-08-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT01602614/Prot_000.pdf
  • Statistical Analysis Plan (2013-05-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT01602614/SAP_001.pdf